CLINICAL TRIAL: NCT05634317
Title: Supporting Family Caregivers of People With Dementia and Identifying an Effective Adaptive Intervention to Reduce Their Depressive Symptoms: a Sequential Multiple Assignment Randomized Trial
Brief Title: Supporting Caregivers of PWD and Identifying an Effective Intervention to Reduce Their Depressive Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Patrick KOR Pui Kin, Assistant Professor, School of nursing, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: TBC
Record Dates: First submitted 2022-10-10; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral activation (Experimental): The SD-BA, consisting of 16 sessions (30 minutes each) twice a week over 8 weeks, will be delivered by the trained instructor through a videoconference mobile app. Participants will be asked to review their daily activity patterns and then choose activity goals and review their successes and areas of improvement. They will also be taught how to fill out the daily monitoring record, which will involve noting down their activities on the day of the session for each hour before the session, and rating the importance and degree of enjoyment associated with each activity.
  Interventions: Behavioral: Smartphone delivered Behavioral activation
- Mindfulness (Active Comparator): A mindfulness instructor will deliver the program through a videoconference mobile app, and include various mindfulness practices (e.g., mindful walking, body scanning) and sharing. To standardize the interventions in this study, the previous approach will be changed from 7 weekly 120-minute sessions to 16 sessions (30 minutes each) twice a week over 8 weeks. The participants will also be encouraged to perform 30 minutes of mindfulness practice every day. All participants will be given an audio (mp3) recording of guided mindfulness activities to enhance their daily practice, and a logbook via a mobile app or in hardcopy (according to their preference) to record the frequency of their self-practice at home and monitor their compliance rate. Our volunteers will provide support via smartphone to answer questions and address difficulties.
  Interventions: Behavioral: Smartphone delivered Mindfulness

INTERVENTIONS:
Behavioral: Smartphone delivered Behavioral activation — Outline:
  Session 0 45-minute psychoeducation on caregiving and depression
  Session 1 Review the present use of time and use the monitoring form
  Session 2 Brain-storm pleasant events and schedule pleasant activities
  Session 3 Review scheduling of events and discuss how to improve
  Session 4 Review modifications and consolidate gains on scheduling
  Session 5 Review present social support and explore new sources of support
  Session 6 Examine communication skills and explore new options
  Session 7 Review new communications and discuss how to improve
  Session 8 Review modification and consolidate gains on support
  Arms: Behavioral activation
Behavioral: Smartphone delivered Mindfulness — Outline:
  Session 0 45-minute psychoeducation on caregiving and depression
  Session 1 The Raisin exercise (eating meditation) and12-min body scan
  Session 2 Exercises on thoughts and feelings 12-min body scan
  Session 3 Exercises focusing on unpleasant experiences, practicing seeing and hearing , sitting meditation, 3-min breathing space, and mindful stretching and breath meditation
  Session 4 Practicing seeing and hearing, mindful communication, 3-min breathing space, and sitting meditation
  Session 5 Mindful walking, 3-min breathing space, and sitting meditation
  Session 6 Sitting meditation, exercises on thoughts and alternative viewpoints, and 3-min breathing space (responsive)
  Session 7 Sitting meditation, activity and mood exercise, identifying habitual emotional reactions to difficulties, and 3-min breathing space (responsive)
  Session 8 12-min body scan, exercise on looking forward, and exercise on preparing for the future
  Arms: Mindfulness

SUMMARY:
Effective clinical management of chronic conditions like depressive symptoms of caregivers actually requires a sequence of interventions, each adapts to responses to prior interventions, and hence multiple intervention decisions throughout the whole careers of dementia caregivers. The main objective of this study is to build the capacity in the community to support the family caregivers of PWD and identify a 2-stage adaptive intervention involving behavioral activation and mindfulness practice to reduce their depressive symptoms using SMART design. A random sample of 272 family caregivers of PWD who meet the clinical criteria of subthreshold depression will be recruited. Participants will be assessed at T1 (baseline assessment); T2 (immediately after the first stage intervention); T3 (immediately after the 2nd stage intervention); T4 (3 months after the 2nd stage intervention); T5 (6 months after the 2nd stage intervention) with various health-related outcomes. The findings will inform us whether the SMART is efficient in identifying an effective adaptive intervention for reducing depressive symptoms. More importantly, will also show us how to alleviate the negative impact of caregiving in the family caregivers.

DETAILED DESCRIPTION:
Aims The main objective of this study is to build the capacity in the community to support the family caregivers of PWD and identify a 2-stage adaptive intervention involving behavioral activation and mindfulness practice to reduce their depressive symptoms using SMART design. Using a sequential multiple randomized trial (SMART), we aim to investigate whether (1) the smartphone-delivered behavioral activation (SD-BA) or smartphone-delivered mindfulness practice (SD- MP) is more effective for reducing depressive symptoms as the first-stage intervention; (2) evaluate whether extending the original first stage intervention with an additional self-efficacy enhancing component or switching to an alternative intervention is more effective in reducing depressive symptoms when participants are not responding to the first stage intervention; (3) evaluate the sequence of the intervention, SD-BA followed by SD-MP or SD-MP followed by SD-BA is more effective in reducing depressive symptoms; and 4) identify which of our four embedded adaptive interventions (SD- BA with booster for responders and (SD-BA for nonresponses; SD-BA with booster for responders and SD-MP for no responders; SD-MY with booster for responders and SD-MP for non-responders; SD-MP with booster for responders and SD-BA for non-responders) is the most effective for reducing depressive symptoms.

Methods A random sample of 272 family caregivers of PWD who meet the clinical criteria of subthreshold depression will be recruited. Participants will be assessed at T1 (baseline assessment); T2 (immediately after the first stage intervention); T3 (immediately after the 2nd stage intervention); T4 (3 months after the 2nd stage intervention); T5 (6 months after the 2nd stage intervention) with various health-related outcomes.

Significance and value The findings will not only inform us whether the SMART is an efficient approach for identifying an effective adaptive intervention for reducing depressive symptoms, but , more importantly will also show us how to alleviate the negative impact of caregiving in the family caregivers.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 or above
2. FC of an individual with a confirmed medical diagnosis of any type of dementia who has been residing in the community;
3. having been providing care for at least 3 months prior to recruitment
4. the presence of mild-to- moderate depressive symptoms (Patient Health Questionnaire-9 (PHQ-9) score 5 to 14).

Exclusion Criteria:

1. having participated in any structured mind-body intervention, cognitive therapy, or structured psychosocial intervention 6 months prior to recruitment
2. having acute psychiatric and medical comorbidities that are potentially life- threatening or would limit the caregivers' participation or adherence (e.g., suicidal ideation, acute psychosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
The 9-item Chinese version of the Patient Health Questionnaire 9 (PHQ-9) | baseline assessment(T1), after the 1 stage (8th week) (T2), after the second stage (16th week)(T3), 3 months after the 2 stage (T4), and 6 months after the 2 stage (T5))
  PHQ-9* is a 9-question instrument to screen for depression. It requires participants to answer their depression experiences over the past 2 weeks.
  Comparisons of changes of the Patient Health Questionnaire 9 will be considered as follows:
  T1 - T2; T1 - T3; T1 - T4; T1 - T5; T2 - T3; T2 - T4; T2-T5 T3 - T4: T3-T5

SECONDARY OUTCOMES:
Perceived caregiving stress (PSS) | baseline assessment(T1), after the 1 stage (8th week) (T2), after the second stage (16th week)(T3), 3 months after the 2 stage (T4), and 6 months after the 2 stage (T5))
  Perceived Stress Scale contains 10 items with 5-point Likert-type scale rating from 0 (never) to 4 (very often). The total score can range from 0 to 40 with higher scores indicating higher perceived stress.
  Comparisons of changes of the perceived caregiving stress will be considered as follows:
  T1 - T2; T1 - T3; T1 - T4; T1 - T5; T2 - T3; T2 - T4; T2-T5 T3 - T4: T3-T5
Positive Aspect of Caregiving scale (PAC) | baseline assessment(T1), after the 1 stage (8th week) (T2), after the second stage (16th week)(T3), 3 months after the 2 stage (T4), and 6 months after the 2 stage (T5))
  The PAC scale demonstrates the acceptable levels of internal consistency Cronbach's alpha 0.85 among the family caregivers of PWD in Hong Kong. Higher scores indicating more positive self-perceptions of caregiving.
  Comparisons of changes of the positive aspect of caregiving scale will be considered as follows:
  T1 - T2; T1 - T3; T1 - T4; T1 - T5; T2 - T3; T2 - T4; T2-T5 T3 - T4: T3-T5
Pittsburgh Sleep Quality Index | baseline assessment(T1), after the 1 stage (8th week) (T2), after the second stage (16th week)(T3), 3 months after the 2 stage (T4), and 6 months after the 2 stage (T5))
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score.
  Comparisons of changes of the Pittsburgh sleep quality index will be considered as follows:
  T1 - T2; T1 - T3; T1 - T4; T1 - T5; T2 - T3; T2 - T4; T2-T5 T3 - T4: T3-T5
The WHOQOL-OLD BREF (HK) | baseline assessment(T1), after the 1 stage (8th week) (T2), after the second stage (16th week)(T3), 3 months after the 2 stage (T4), and 6 months after the 2 stage (T5))
  The WHOQOL-OLD BREF (HK) comprised 28 items and each item is rated on a 5-point Likert-type scale that ranged from 1 (very dissatisfied) to 5 (very satisfied), with a higher score indicating a better QoL.
  Comparisons of changes of the WHOQOL-OLD BREF (HK) will be considered as follows:
  T1 - T2; T1 - T3; T1 - T4; T1 - T5; T2 - T3; T2 - T4; T2-T5 T3 - T4: T3-T5

OTHER OUTCOMES:
Five Facets Mindfulness Questionnaire-Short Form | baseline assessment(T1), after the 1 stage (8th week) (T2), after the second stage (16th week)(T3), 3 months after the 2 stage (T4), and 6 months after the 2 stage (T5))
  Caregivers' level of mindfulness will be measured as the process indicator by using the Five Facets Mindfulness Questionnaire Short Form. It is a self-report questionnaire measuring the five facets of mindfulness which includes observing, describing, acting with awareness, non-judging of inner and non-reactivity to inner experience (e.g., "I'm good at finding words to describe my feelings"). The total score ranges from 20 to 100 and the higher the score, the higher level of mindfulness.
  Comparisons of changes of the five facets mindfulness questionnaire-short form will be considered as follows:
  T1 - T2; T1 - T3; T1 - T4; T1 - T5; T2 - T3; T2 - T4; T2-T5 T3 - T4: T3-T5

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic Univeristy, Hong Kong, Hong Kong

REFERENCES:
- [Background] Organization WH. Dementia: key facts. Retrieved March. 2019;31:2020.
- [Background] Elderly Health Service DoHHK. Dementia. In: Health Do, editor. Hong Kong2016.
- [Background] Romero-Moreno R, Losada A, Marquez-Gonzalez M, Mausbach BT. Stressors and anxiety in dementia caregiving: multiple mediation analysis of rumination, experiential avoidance, and leisure. Int Psychogeriatr. 2016 Nov;28(11):1835-1844. doi: 10.1017/S1041610216001009. Epub 2016 Jul 26. PMID 27457894
- [Background] Anand KS, Dhikav V, Sachdeva A, Mishra P. Perceived caregiver stress in Alzheimer's disease and mild cognitive impairment: A case control study. Ann Indian Acad Neurol. 2016 Jan-Mar;19(1):58-62. doi: 10.4103/0972-2327.167695. PMID 27011630
- [Background] Afram B, Stephan A, Verbeek H, Bleijlevens MH, Suhonen R, Sutcliffe C, Raamat K, Cabrera E, Soto ME, Hallberg IR, Meyer G, Hamers JP; RightTimePlaceCare Consortium. Reasons for institutionalization of people with dementia: informal caregiver reports from 8 European countries. J Am Med Dir Assoc. 2014 Feb;15(2):108-16. doi: 10.1016/j.jamda.2013.09.012. Epub 2013 Nov 12. PMID 24238605
- [Background] Zhu CW, Scarmeas N, Ornstein K, Albert M, Brandt J, Blacker D, Sano M, Stern Y. Health-care use and cost in dementia caregivers: Longitudinal results from the Predictors Caregiver Study. Alzheimers Dement. 2015 Apr;11(4):444-54. doi: 10.1016/j.jalz.2013.12.018. Epub 2014 Mar 15. PMID 24637299
- [Background] O'Dwyer ST, Moyle W, Zimmer-Gembeck M, De Leo D. Suicidal ideation in family carers of people with dementia. Aging Ment Health. 2016;20(2):222-30. doi: 10.1080/13607863.2015.1063109. Epub 2015 Jul 10. PMID 26161825
- [Background] Zabihi S, Lemmel FK, Orgeta V. Behavioural Activation for Depression in Informal Caregivers: A Systematic Review and Meta-Analysis of Randomised Controlled Clinical Trials. J Affect Disord. 2020 Sep 1;274:1173-1183. doi: 10.1016/j.jad.2020.03.124. Epub 2020 Apr 29. PMID 32663948
- [Background] Cheng ST, Li KK, Losada A, Zhang F, Au A, Thompson LW, Gallagher-Thompson D. The effectiveness of nonpharmacological interventions for informal dementia caregivers: An updated systematic review and meta-analysis. Psychol Aging. 2020 Feb;35(1):55-77. doi: 10.1037/pag0000401. PMID 31985249
- [Background] Walter E, Pinquart M. How Effective Are Dementia Caregiver Interventions? An Updated Comprehensive Meta-Analysis. Gerontologist. 2020 Nov 23;60(8):609-619. doi: 10.1093/geront/gnz118. PMID 33226434
- [Background] Richards DA, Ekers D, McMillan D, Taylor RS, Byford S, Warren FC, Barrett B, Farrand PA, Gilbody S, Kuyken W, O'Mahen H, Watkins ER, Wright KA, Hollon SD, Reed N, Rhodes S, Fletcher E, Finning K. Cost and Outcome of Behavioural Activation versus Cognitive Behavioural Therapy for Depression (COBRA): a randomised, controlled, non-inferiority trial. Lancet. 2016 Aug 27;388(10047):871-80. doi: 10.1016/S0140-6736(16)31140-0. Epub 2016 Jul 23. PMID 27461440
- [Background] Xu XY, Kwan RYC, Leung AYM. Behavioural activation for family dementia caregivers: A systematic review and meta-analysis. Geriatr Nurs. 2020 Sep-Oct;41(5):544-552. doi: 10.1016/j.gerinurse.2020.02.003. Epub 2020 Mar 3. PMID 32143964
- [Background] Au A, Gallagher-Thompson D, Wong MK, Leung J, Chan WC, Chan CC, Lu HJ, Lai MK, Chan K. Behavioral activation for dementia caregivers: scheduling pleasant events and enhancing communications. Clin Interv Aging. 2015 Mar 26;10:611-9. doi: 10.2147/CIA.S72348. eCollection 2015. PMID 25848237
- [Background] Au A, Yip HM, Lai S, Ngai S, Cheng ST, Losada A, Thompson L, Gallagher-Thompson D. Telephone-based behavioral activation intervention for dementia family caregivers: Outcomes and mediation effect of a randomized controlled trial. Patient Educ Couns. 2019 Nov;102(11):2049-2059. doi: 10.1016/j.pec.2019.06.009. Epub 2019 Jun 26. PMID 31279613
- [Background] Kor PPK, Chien WT, Liu JYW, Lai CKY. Mindfulness-Based Intervention for Stress Reduction of Family Caregivers of People with Dementia: A Systematic Review and Meta-Analysis. Mindfulness. 2018;9(1):7-22.
- [Background] Kor PPK, Liu JYW, Chien WT. Effects of a modified mindfulness-based cognitive therapy for family caregivers of people with dementia: A pilot randomized controlled trial. Int J Nurs Stud. 2019 Oct;98:107-117. doi: 10.1016/j.ijnurstu.2019.02.020. Epub 2019 Mar 8. PMID 30922609
- [Background] Cheung DSK, Kor PPK, Jones C, Davies N, Moyle W, Chien WT, Yip ALK, Chambers S, Yu CTK, Lai CKY. The Use of Modified Mindfulness-Based Stress Reduction and Mindfulness-Based Cognitive Therapy Program for Family Caregivers of People Living with Dementia: A Feasibility Study. Asian Nurs Res (Korean Soc Nurs Sci). 2020 Oct;14(4):221-230. doi: 10.1016/j.anr.2020.08.009. Epub 2020 Sep 12. PMID 32931996
- [Background] Liu Y, Kim K, Zarit SH. Health trajectories of family caregivers: associations with care transitions and adult day service use. J Aging Health. 2015 Jun;27(4):686-710. doi: 10.1177/0898264314555319. Epub 2014 Oct 27. PMID 25348275
- [Background] Kor PPK, Liu JYW, Chien WT. Effects of a Modified Mindfulness-Based Cognitive Therapy for Family Caregivers of People With Dementia: A Randomized Clinical Trial. Gerontologist. 2021 Aug 13;61(6):977-990. doi: 10.1093/geront/gnaa125. PMID 32886746
- [Background] Almirall D, Compton SN, Gunlicks-Stoessel M, Duan N, Murphy SA. Designing a pilot sequential multiple assignment randomized trial for developing an adaptive treatment strategy. Stat Med. 2012 Jul 30;31(17):1887-902. doi: 10.1002/sim.4512. Epub 2012 Mar 22. PMID 22438190
- [Background] Jiang D, Warner LM, Chong AM, Li T, Wolff JK, Chou KL. Promoting Volunteering Among Older Adults in Hong Kong: A Randomized Controlled Trial. Gerontologist. 2020 Jul 15;60(5):968-977. doi: 10.1093/geront/gnz076. PMID 31228197
- [Background] Oetting A, Levy J, Weiss R, Murphy S. Causality and psychopathology: Finding the determinants of disorders and their cures. Shrout, P. 2007.
- [Background] Bellg AJ, Borrelli B, Resnick B, Hecht J, Minicucci DS, Ory M, Ogedegbe G, Orwig D, Ernst D, Czajkowski S; Treatment Fidelity Workgroup of the NIH Behavior Change Consortium. Enhancing treatment fidelity in health behavior change studies: best practices and recommendations from the NIH Behavior Change Consortium. Health Psychol. 2004 Sep;23(5):443-51. doi: 10.1037/0278-6133.23.5.443. PMID 15367063
- [Background] Brown EL, Ruggiano N, Li J, Clarke PJ, Kay ES, Hristidis V. Smartphone-Based Health Technologies for Dementia Care: Opportunities, Challenges, and Current Practices. J Appl Gerontol. 2019 Jan;38(1):73-91. doi: 10.1177/0733464817723088. Epub 2017 Aug 4. PMID 28774215
- [Background] Mak WW, Tong AC, Yip SY, Lui WW, Chio FH, Chan AT, Wong CC. Efficacy and Moderation of Mobile App-Based Programs for Mindfulness-Based Training, Self-Compassion Training, and Cognitive Behavioral Psychoeducation on Mental Health: Randomized Controlled Noninferiority Trial. JMIR Ment Health. 2018 Oct 11;5(4):e60. doi: 10.2196/mental.8597. PMID 30309837
- [Background] Choi NG, Caamano J, Vences K, Marti CN, Kunik ME. Acceptability and effects of tele-delivered behavioral activation for depression in low-income homebound older adults: in their own words. Aging Ment Health. 2021 Oct;25(10):1803-1810. doi: 10.1080/13607863.2020.1783516. Epub 2020 Jul 22. PMID 32693614
- [Background] Segal ZV, Williams JMG, Teasdale JD. Mindfulness-based cognitive therapy for depression : a new approach to preventing relapse. New York: New York : Guilford Press; 2002.
- [Background] Yu X, Tam WW, Wong PT, Lam TH, Stewart SM. The Patient Health Questionnaire-9 for measuring depressive symptoms among the general population in Hong Kong. Compr Psychiatry. 2012 Jan;53(1):95-102. doi: 10.1016/j.comppsych.2010.11.002. Epub 2010 Dec 28. PMID 21193179
- [Background] Leung DY, Lam TH, Chan SS. Three versions of Perceived Stress Scale: validation in a sample of Chinese cardiac patients who smoke. BMC Public Health. 2010 Aug 25;10:513. doi: 10.1186/1471-2458-10-513. PMID 20735860
- [Background] Lou VW, Lau BH, Cheung KS. Positive aspects of caregiving (PAC): scale validation among Chinese dementia caregivers (CG). Arch Gerontol Geriatr. 2015 Mar-Apr;60(2):299-306. doi: 10.1016/j.archger.2014.10.019. Epub 2014 Nov 7. PMID 25488014
- [Background] Chong AML, Cheung C-k. Factor structure of a Cantonese-version Pittsburgh Sleep Quality Index. Sleep and Biological Rhythms. 2012;10(2):118-25.
- [Background] Zeng Q-Z, He Y-L, Liu H, Miao J-M, Chen J-X, Xu H-N, et al. Reliability and validity of Chinese version of the Generalized Anxiety Disorder 7-item (GAD-7) scale in screening anxiety disorders in outpatients from traditional Chinese internal department. [Reliability and validity of Chinese version of the Generalized Anxiety Disorder 7-item (GAD-7) scale in screening anxiety disorders in outpatients from traditional Chinese internal department.]. Chinese Mental Health Journal. 2013;27(3):163-8.
- [Background] Wong ELY, Ramos-Goni JM, Cheung AWL, Wong AYK, Rivero-Arias O. Assessing the Use of a Feedback Module to Model EQ-5D-5L Health States Values in Hong Kong. Patient. 2018 Apr;11(2):235-247. doi: 10.1007/s40271-017-0278-0. PMID 29019161
- [Background] Hou J, Wong SY, Lo HH, Mak WW, Ma HS. Validation of a Chinese version of the Five Facet Mindfulness Questionnaire in Hong Kong and development of a short form. Assessment. 2014 Jun;21(3):363-71. doi: 10.1177/1073191113485121. Epub 2013 Apr 16. PMID 23596271
- [Background] Verbeke G. Linear mixed models for longitudinal data. Linear mixed models in practice: Springer; 1997. p. 63-153.
- [Background] Nahum-Shani I, Qian M, Almirall D, Pelham WE, Gnagy B, Fabiano GA, Waxmonsky JG, Yu J, Murphy SA. Experimental design and primary data analysis methods for comparing adaptive interventions. Psychol Methods. 2012 Dec;17(4):457-477. doi: 10.1037/a0029372. Epub 2012 Oct 1. PMID 23025433
- [Background] Greenglass ER, Fiksenbaum L. Proactive coping, positive affect, and well-being: Testing for mediation using path analysis. European psychologist. 2009;14(1):29-39.
- [Background] Glick HA, Doshi JA, Sonnad SS, Polsky D. Economic evaluation in clinical trials: OUP Oxford; 2014.
- [Derived] Kor PPK, Chou KL, Zarit SH, Gallagher D, Galante J, Wong SYS, Cheung DSK, Leung AYM, Chu LW. Sequential multiple assignment randomised controlled trial protocol for developing an adaptive intervention to improve depressive symptoms among family caregivers of people with dementia. BMJ Open. 2023 Sep 6;13(9):e072410. doi: 10.1136/bmjopen-2023-072410. PMID 37673447